CLINICAL TRIAL: NCT06941584
Title: Analysis of the Role of AIRE in Autoimmune Neurological Diseases Associated With Autoantibodies
Acronym: NAD-AIRE
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Other Study IDs: 6449
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-03

CONDITIONS: AIRE Deficiency
Keywords: AIRE gene mutation; Myasthenia gravis; Neuromyelitis Optica Spectrum Disorder; Acquired neuromyotonia; Autoimmune encephalitis; Thymic central tolerance; HLA haplotype
MeSH Terms: conditions — Polyendocrinopathies, Autoimmune; Myasthenia Gravis; Neuromyelitis Optica; Isaacs Syndrome; Autoimmune Diseases of the Nervous System | interventions — Alleles

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — AIRE single gene sequencing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First cohort - Patients with diagnosis of a neurological autoimmune disease: For the first cohort, the inclusion criteria were:
  * Patients diagnosed with NMOSD associated with AQP4 autoantibodies who meet the 2015 diagnostic criteria and have at least one of the listed autoimmune comorbidities.
  * Patients diagnosed with myasthenia gravis associated with AChR autoantibodies who also have another autoimmune comorbidity from the list.
  * Patients diagnosed with autoimmune encephalitis who are positive for LGI1 and CASPR2 autoantibodies and have at least one additional autoimmune comorbidity.
  The only exclusion criterion was the presence of untreated thymoma or a history of thymoma.
  Interventions: Genetic: AIRE single gene sequencing; Genetic: Molecular typing of HLA class I and II alleles
- Second cohort - Patients with AIRE mutations: The second cohort included adults with dominant pathogenic AIRE mutations or homozygous AIRE mutations.
  Interventions: Diagnostic Test: Test for AQP4, AChR, LGI1, and CASPR2 autoantibodies using cell-based assay; Genetic: Molecular typing of HLA class I and II alleles

INTERVENTIONS:
Diagnostic Test: Test for AQP4, AChR, LGI1, and CASPR2 autoantibodies using cell-based assay — To evaluate the prevalence of specific autoantibodies (AQP4, AChR, LGI1, and CASPR2) in the population of patients carrying AIRE mutations (second cohort)
  Groups: Second cohort - Patients with AIRE mutations
Genetic: AIRE single gene sequencing — To assess the prevalence of AIRE gene mutations in patients with NMOSD associated with AQP4 autoantibodies, myasthenia gravis (MG) associated with AChR autoantibodies, acquired neuromyotonia, and autoimmune encephalitis associated with CASPR2 and LGI1 autoantibodies (first cohort)
  Groups: First cohort - Patients with diagnosis of a neurological autoimmune disease
Genetic: Molecular typing of HLA class I and II alleles — To assess the HLA haplotypes of class I and II by comparing patients with and without AIRE mutations, as well as those with and without autoimmune neurological diseases

SUMMARY:
Studying genetic predisposition in autoimmune neurological diseases could help improve diagnostic accuracy and offer new treatment possibilities

DETAILED DESCRIPTION:
Autoimmune diseases involving the nervous system include conditions affecting both the central nervous system (CNS)-such as neuromyelitis optica spectrum disorder (NMOSD) and autoimmune encephalitis-and the peripheral nervous system, as exemplified by myasthenia gravis (MG), which targets the neuromuscular junction. Although these disorders present with distinct clinical features, they share a common immunopathogenic hallmark: the presence of pathogenic autoantibodies directed against neural or neuromuscular antigens.

While the mechanisms underlying the production of these autoantibodies remain only partially understood, increasing evidence points to defects in immune tolerance as key contributors to disease onset. In MG, in particular, the thymus is directly implicated in the disease process, with thymic follicular hyperplasia observed in early-onset forms and thymoma present in a significant subset of patients. Notably, reduced expression of the autoimmune regulator gene (AIRE) has been demonstrated in thymomas associated with MG, suggesting a failure of central immune tolerance in the pathogenesis of this condition.

Additionally, other autoimmune diseases of the CNS, such as neuromyelitis optica (NMOSD) and autoimmune encephalitis, have been associated with the contribution of peripheral tolerance in promoting the onset and maintenance of autoimmunity.

However, several studies suggest that the thymic escape of autoreactive T cells is an important pathophysiological mechanism in CNS autoimmune diseases mediated by autoantibodies. In animal models, thymic negative selection is a critical factor in determining susceptibility and severity of CNS inflammation. There is also indirect clinical data suggesting that thymic function is important in human CNS autoimmune diseases. In particular, the association between thymoma and paraneoplastic encephalitis-such as in the case of encephalitis associated with voltage-gated potassium channel (VGKC) complex antibodies (CASPR2 and LGI1)-highlights the involvement of thymic tolerance in these diseases.

Thymic central tolerance is orchestrated by thymic epithelial cells (TECs), the most abundant stromal cells, located in the cortical (cTEC) and medullary (mTEC) regions.

As known, HLA plays a crucial role in the selection of T-cells within the thymus. In the initial phase, only those T-cells whose TCRs bind to HLA molecules expressed by epithelial cells in the thymic cortex are positively selected, while the others undergo apoptosis. Immature thymocytes co-express both CD4 and CD8, but if their TCR preferentially recognizes class I HLA, they downregulate CD4 and upregulate CD8; conversely, if they recognize class II HLA, the opposite occurs.

The T-cells then migrate to the thymic medulla, where a broad array of self-peptides bound to HLA I and II are presented. At this stage, thymocytes that form high-affinity interactions with these self-peptides are eliminated, a process that helps suppress autoimmunity and foster self-tolerance. Several mechanisms have been proposed that link HLA to disease, often involving the failure of thymic negative selection due to disturbances in the TCR-peptide-HLA interaction.

The ectopic expression of thousands of genes, including tissue-specific antigens (TRA) by mTECs, is crucial for eliminating T cells that bind to these antigens. The recognition of autoantigens in the thymus is facilitated by multigenic transcription factors, such as AIRE (autoimmune regulator), expressed in the thymic medulla. AIRE plays a crucial role in inducing the expression of peripheral antigens in the thymus, enabling the elimination of autoreactive T cells through negative selection.

The congenital loss of AIRE function leads to autoimmune polyglandular syndrome type 1 (APS1). This condition is characterized by a combination of Addison's disease, hypoparathyroidism, chronic mucocutaneous candidiasis, and several other autoimmune diseases caused by the presentation of a limited repertoire of autoantigens by mTECs, compromising the removal of autoreactive T cells. The manifestations of APS1 underscore the crucial role of AIRE in the presentation of autoantigens in the thymus and in building thymic tolerance.

Despite the central role of the AIRE gene in mediating thymic tolerance, its contribution to the pathogenesis of autoimmune neurological diseases remains largely unexplored. While previous research has focused on peripheral tolerance mechanisms, few studies have investigated how AIRE dysfunction might affect the presentation of key neural autoantigens-such as AQP4, AChR, LGI1, and CASPR2-within medullary thymic epithelial cells (mTECs).

Notably, no systematic screening for pathogenic antibodies has been conducted in patients with AIRE mutations, and the role of AIRE gene variants in patients with NMOSD, myasthenia gravis, or autoimmune encephalitis remains undefined.

Another important factor contributing to susceptibility to autoimmune diseases is HLA typing. Several studies have demonstrated that specific HLA haplotypes are associated with an increased risk of developing autoimmune neurological diseases. In particular, NMOSD has been associated with the HLA-DRB1*03:01 haplotype, which seems to be a significant risk factor in anti-AQP4 positive patients (Zéphir et al., 2009). Similarly, myasthenia gravis is strongly correlated with HLA-DR3, especially in patients with early-onset disease (Berrih-Aknin, 2017). Moreover, autoimmune encephalitis associated with autoantibodies against LGI1 and CASPR2 shows a significant association with HLA-DRB1*07:01, suggesting a crucial role for HLA in antigen presentation and the development of neurological autoimmunity (Kim et al., 2017; van Sonderen et al., 2017).

The aim of this study is to explore the role of the AIRE gene in the pathogenesis of autoimmune neurological diseases and investigate how specific HLA haplotypes may predispose individuals to develop these conditions.

Our hypothesis is that alterations in AIRE expression and dysfunctions in central tolerance may contribute to the development of neurological autoimmunity, especially in individuals with certain high-risk HLA haplotypes.

ELIGIBILITY:
Inclusion Criteria:

For the first cohort, the inclusion criteria were:

* Patients diagnosed with NMOSD associated with AQP4 autoantibodies who meet the 2015 diagnostic criteria and have at least one of the listed autoimmune comorbidities.
* Patients diagnosed with myasthenia gravis associated with AChR autoantibodies who also have another autoimmune comorbidity from the list.
* Patients diagnosed with autoimmune encephalitis who are positive for LGI1 and CASPR2 autoantibodies and have at least one additional autoimmune comorbidity.

The second cohort included adults with dominant pathogenic AIRE mutations or homozygous AIRE mutations.

Exclusion Criteria:

The presence of untreated thymoma or a history of thymoma.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The first cohort includes adults (aged over 18 years) diagnosed with autoimmune neurological diseases, such as NMOSD, myasthenia gravis, and autoimmune encephalitis, as well as patients with at least one of the following autoimmune comorbidities: systemic lupus erythematosus, Sjögren's syndrome, rheumatoid arthritis or type 1 diabetes mellitus.
  The second cohort consists of adults (aged over 18 years) with dominant pathogenic mutations in the AIRE gene, as well as patients with homozygous mutations in the same gene.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2027-01-06 (Estimated); Study Completion 2027-01-06 (Estimated)

PRIMARY OUTCOMES:
The role of AIRE in neurological autoimmune diseases | 36 months
  To assess the prevalence of AIRE gene mutations in patients with NMOSD associated with AQP4 autoantibodies, myasthenia gravis (MG) associated with AChR autoantibodies, acquired neuromyotonia, and autoimmune encephalitis associated with CASPR2 and LGI1 autoantibodies

SECONDARY OUTCOMES:
The prevalence of specific autoantibodies (AQP4, AChR, LGI1, CASPR2) in patients carrying AIRE mutations | 36 months
  To evaluate the prevalence of specific autoantibodies (AQP4, AChR, LGI1, and CASPR2) in the population of patients carrying AIRE mutations
The synergy between AIRE gene mutations and HLA haplotype in patients with autoimmune neurological diseases | 36 months
  assess the HLA haplotypes of class I and II by comparing patients with and without AIRE mutations, as well as those with and without autoimmune neurological diseases

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Iorio, MD, Principal Investigator — Dipartimento di Neurologia - Policlinico Fondazione Agostino Gemelli
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, IRCSS Roma, Roma, Italy